CLINICAL TRIAL: NCT00451594
Title: A Randomized Controlled Multicentre Trial of High Dose Dexamethasone Versus Conventional Dose Prednisolone for Adults With Untreated Idiopathic Thrombocytopenic Purpura
Brief Title: High Dose Dexamethasone Vs. Conventional Dose Prednisolone in Adult ITP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: COSAH, Cooperative Study Group A for Hematology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-009
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone; Absorptiometry, Photon; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dexamethasone — Pulse high dose dexamethasone (Arm 1)
  1. Patients will receive 40 mg of oral dexamethasone daily for four consecutive days.
  2. Other treatments should be considered if there was a platelet count of 30X109/L or less by day 14
  3. If the patient had a platelet count of more than 30X109/L after four days of dexamethasone treatment, no further treatment will be given.
  4. If the platelet count drops below 30X109/L within the first 6 months, another four-day course of dexamethasone will be given, followed by 15 mg of prednisone daily, with gradual tapering.
  5. Patients whose platelet counts can not be maintained at 30X109/L will be offered other treatments.
  Other Names: Dexa
Drug: Prednisolone — Conventional dose prednisone (Arm 2)
  1. Prednisone, 1 mg/kg is started at diagnosis. If the platelet count is more than 100X109/L, the dose should be used for 4 weeks minimally and then tapered by 10 mg/1 wk until the dose reaches 0.5 mg/kg of body weight and by 5 mg/1 wk thereafter. (Ann Intern Med 1997, 126, 307-14). If the platelet count is between 30X109/L and 100X109/L, prednisone 1 mg/kg should be used for 8 weeks maximally and then tapered by 10 mg/2 wk until the dose reaches 0.5 mg/kg of body weight and by 5 mg/2 wk thereafter.
  2. Guideline of prednisone tapering Duration of prednisone treatment: 3-6 months
  Other Names: PD

SUMMARY:
To determine the long term effects of pulse high dose dexamethasone and conventional dose prednisolone in treatment of adult patients with ITP.

DETAILED DESCRIPTION:
Patients will be randomized to one of two study arms:

dexamethasone 40 mg po daily for 4 consecutive days. If the platelet count drops below 30X109/L after response within 6 months, another four-day course of dexamethasone will be given, followed by 15 mg of prednisone daily, with gradual tapering (Arm 1).

Prednisone 1 mg/kg po daily for 4-8 weeks, the drug is then decreased slowly over another few weeks (Arm 2).

ELIGIBILITY:
Inclusion Criteria :

* a true thrombocytopenia on blood smear
* adequate megakaryopoiesis on bone marrow examination
* the absence of clinically apparent associated conditions or cause of thrombocytopenia
* Age over 16 years
* A platelet count of less than 30x109/L

Exclusion criteria :

* previous treatment for ITP.
* other causes of thrombocytopenia such as HIV infection, lymphproliferative disease, liver disease, or definite SLE.
* Patients with life threatening bleeding and pregnant women should be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2005-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
response rate and platelet count | 6 years
  Endpoint definitions and criteria for evaluation: This study is designed to compare the effectiveness of high dose dexamethasone with conventional dose prednisone for patient with ITP. The effectiveness will be evaluated in terms of response rate and platelet count at 6 months after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sung Hwa Bae, professor, Principal Investigator — Daegu Catholic Univertity Hospital, ROK; Jung-Hee Lee, professor, Principal Investigator — Asan Medical Center, ROK
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- See also: A RANDOMIZED CONTROLLED MULTICENTER TRIAL OF HIGH DOSE DEXAMETHASONE VERSUS CONVENTIONAL DOSE PREDNISONE FOR ADULTS WITH UNTREATED IDIOPATHIC THROMBOCYTOPENIC PURPURA — http://www.google.co.kr